CLINICAL TRIAL: NCT04129333
Title: HYPIC Hypnosis for Procedural Pain in the Intensive Care Unit
Acronym: HYPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35RC18_8853_HYPIC; 2019-A01775-52 (Other: ID RCB)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Invasive Procedure
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Multicenter prospective national, controlled, randomized, superiority study, open-label with blind evaluation, on 2 parallel groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental): A hypnosis group with standard care during the invasive procedure according to the usual practice of the care team and setting up a hypnotic accompaniment by an nurse trained beforehand and dedicated throughout the gesture. The hypnosis session will end at the same time as the invasive procedure.
  Interventions: Other: Hypnosis
- Control group (Placebo Comparator): A control group with standard care during the invasive procedure according to the usual practice of the care team.
  Interventions: Other: No hypnosis

INTERVENTIONS:
Other: Hypnosis — The hypnosis session :
  * Creation of the therapist-patient link
  * Choice of a theme and the preferred sensory channel by the patient
  * Collection of the theme chosen by the patient
  * Orientation in the here and now.
  * Induction
  * Realization of the gesture and hypnosis
  * At the end of the procedure, reassociation of the patient in the here and now
  Arms: Hypnosis group
Other: No hypnosis — No hypnosis
  Arms: Control group

SUMMARY:
Procedural pain in resuscitation is common in the conscious patient. However, analgesia and sedation may be impossible because of the acute pathology leading to resuscitation, comorbidities or the urgency of the invasive procedure. In addition, the use of analgesics and sedatives is responsible for adverse effects. In this context, hypnosis appears to be an additional analgesic tool that would reduce the consumption of analgesics and sedatives and thus reduce their side effects.

ELIGIBILITY:
Inclusion Criteria:

* Major patient admitted to intensive care
* Glasgow score = 15
* Necessity during the stay of making an invasive gesture among:
* Thoracic drainage
* Placement of a central venous catheter or a Swan-Ganz catheter
* Establishment of a dialysis catheter
* Introduction of an invasive arterial catheter
* Patient giving free, informed and written consent
* Patient affiliated to a social security scheme

Non inclusion Criteria:

* Procedure to be carried out in extreme urgency
* Confusional state making hypnosis impossible, evaluated by CAM-ICU (Confusion Assessment Method for the Intensive Care Unit)
* Decompensated psychiatric illness
* Patient sedated or intravenous analgesia continued at the time of the procedure
* Patient intubated
* Patient with a contraindication to sedation or analgesia at the time of the procedure
* Patient receiving topical anesthesia before the start of the procedure
* Major person subject to legal protection (court bail, curator, guardianship) or deprived of liberty
* Patient already included in the study during the completion of a previous invasive procedure
* Patient participating in a research involving an interventional human person (category 1) on an analgesic / sedative drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Immediately after the end of the invasive procedure (Hour 0)
  Oral assessment scale (0 : no pain - 10 : maximal pain)

SECONDARY OUTCOMES:
Pain assessment | The first hour after the end of the procedure (Hour 1)
  Oral assessment scale (0 : no pain - 10 : maximal pain)
Morphine equivalent dose | Immediately after the end of the invasive procedure (H0) and the first hour after the end of the procedure (H1)
  Cumulative use of morphine-morphine analgesics in morphine equivalent during the procedure and the first hour after the end of the procedure (H1)
Sedatives dose | Immediately after the end of the invasive procedure (Hour 0) and the first hour after the end of the procedure (Hour 1)
  Cumulative use of sedatives during the procedure and the first hour after the end of the procedure (H1)
Local Anesthesia dose | Immediately after the end of the invasive procedure (Hour 0)
  Consumption of local anesthesia during the invasive procedure
Comfort scale | Immediately after the end of the invasive procedure (H0) and the first hour after the end of the procedure (H1)
  Comfort measured by the numerical comfort scale (0 no comfort - 10 most comfortable situation imaginable)
Anxiety | Immediately after the end of the invasive procedure (Hour 0) and the first hour after the end of the procedure (Hour 1)
  Patient anxiety measured by the numerical anxiety scale (0 no anxiety - 10 greatest anxiety imaginable) .
Duration | Immediately after the end of the invasive procedure (Hour 0)
  Duration of the invasive procedure including the period of hypnosis
Number of attempts and failures of the procedure | The first hour after the end of the procedure (Hour 1)
  Number of attempts and failures of the procedure
Adverse events | The first hour after the end of the procedure (Hour 1)
  Number of adverse events occurring during the procedure (hematoma, failure to pose, ...)
Nurse stress | Immediately after the end of the invasive procedure (Hour 0)
  Stress of the nurse in charge of the patient quantified by a numerical scale of evaluation (0 no stress - 10 greatest stress imaginable)
Length of stay in intensive care unit | Day 28
  Length of stay in intensive care unit, measured until D28

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Saint-Brieuc Hospital, Saint-Brieuc, Brittany Region
  - Rennes University Hospital, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maamar A, Faleur C, Pedrono K, Adeux MP, Anne M, Verdes A, Fillatre P, Debarre M, Mercier N, Revest M, Massart N, Poilvet N, Terzi N, Tadie JM, Gacouin A, Laviolle B. Hypnosis for unplanned procedural pain in the intensive care unit: the HYPIC randomized clinical trial. Crit Care. 2025 Jul 18;29(1):312. doi: 10.1186/s13054-025-05563-9. PMID 40682163